CLINICAL TRIAL: NCT03673878
Title: Study on the Prevalence of a Localized or Diffuse Pruritus in a Population With One or Several, Primitive or Secondary, Brain Tumor(s)
Brief Title: Prevalence of a Localized or Diffuse Pruritus in a Population With One or Several, Primitive or Secondary, Brain Tumor(s)
Acronym: PRURI-C
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC18.0155
Record Dates: First submitted 2018-08-14; First posted 2018-09-17 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Pruritus; Brain Tumor
MeSH Terms: conditions — Pruritus; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association between the presence of pruritus, especially centrofacial, and the presence of a brain tumor is a widespread notion in the medical community but based on a single publication by Andreev et al. in the British Journal of Dermatology published in 1975. No other study has studied this association with a rigorous methodology. The aim of this study is to evaluate the prevalence of pruritus in patients with one or more primary or secondary brain tumor(s), benign(s) or malignant(s).

DETAILED DESCRIPTION:
* Monocentric prospective observational study
* On the inclusion period
* Patients who are seen in radiotherapy consultation and / or department of neurosurgery
* Complying with the inclusion criteria, not falling within the exclusion criteria
* Re-reading of cerebral MRI (cMRI) with precision on the location(s) of the brain tumor(s) according to a predefined anatomic descriptive diagram
* Complete the questionnaire by a dermatologist (characteristics of pruritus, brain lesion(s), characteristics of the population)

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Diagnosis of benign or malignant brain tumor, primary or secondary.
* Accepted non-opposition
* Realization of a cerebral MRI (cMRI)

Exclusion criteria:

* Age < 18 years
* Absence of cerebral imaging of the cMRI type
* Absence of non opposition
* Realization of a treatment modifying the brain structure (radiotherapy / surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who are seen in radiotherapy consultation and / or hospitalization of neurosurgery Fulfilling the inclusion criteria, not falling within the exclusion criteria Presence of itching for more than 1 week in a patient with one or more brain tumor(s), primary or secondary, benign(s) or malignant(s).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Presence of itching for more than 1 week in a patient with one or more brain tumor(s), primary or secondary, benign(s) or malignant(s). | 1 year
  Presence of itching for more than 1 week in a patient with one or more brain tumor(s), primary or secondary, benign(s) or malignant(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de dermatologie, CHRU BREST, Brest, France